CLINICAL TRIAL: NCT02505919
Title: A Prospective Multicenter Randomized Blinded Study Comparing Aquablation of the Prostate With the AQUABEAM System and TURP for the Treatment of LUTS
Brief Title: Waterjet Ablation Therapy for Endoscopic Resection of Prostate Tissue (WATER)
Acronym: WATER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PROCEPT BioRobotics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TP0038
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Results first posted 2020-04-08 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
Keywords: Lower Urinary Tract Symptoms (LUTS)
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: All study subjects and the study site follow-up team are blinded to the assigned treatment until the year 3 follow-up.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): AQUABEAM System
  Interventions: Device: AQUABEAM System
- Active Comparator (Active Comparator): Transurethral Resection of the Prostate (TURP)
  Interventions: Procedure: Transurethral Resection of the Prostate (TURP)

INTERVENTIONS:
Device: AQUABEAM System — The AQUABEAM system, a personalized image-guided tissue removal system, utilizes proprietary heat-free high-velocity waterjet technology to resect and remove prostate tissue.
  Arms: Treatment
Procedure: Transurethral Resection of the Prostate (TURP) — Transurethral resection of the prostate (TURP) is a type of prostate surgery done to relieve moderate to severe urinary symptoms caused by an enlarged prostate, a condition known as benign prostatic hyperplasia (BPH)
  Arms: Active Comparator

SUMMARY:
A prospective multicenter randomized blinded study comparing Aquablation of the prostate with the AQUABEAM System and TURP for the treatment of Lower Urinary Tract Symptoms (LUTS). The primary endpoints for safety and effectiveness were measured at 3 and 6 months, respectively, and subjects were followed out to 5 years to collect long-term clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Subject has diagnosis of lower urinary tract symptoms due to benign prostatic enlargement causing bladder outlet obstruction.
* Age from 45 to 80 years.
* Subject has medical record documentation of a prostate volume between 30mL and 80mL (inclusive) by transrectal ultrasound (TRUS). (If TRUS testing documentation is available from less than 180 days prior to the informed consent date and the prostate volume is between 30mL and 80mL, it may be used for the inclusion/exclusion criteria.)
* Subject has an International Prostate Symptom Score (IPSS) score greater than or equal to 12 measured at the baseline visit.
* Subject has medical record documentation of a maximum urinary flow rate (Qmax) less than 15mL/s. (If uroflow testing documentation is available within 90 days prior to the informed consent date, and the sample is greater than or equal to 125mL, and the Qmax is less than 15mL/s it may be used for the inclusion/exclusion criteria.)
* Subject has a serum creatinine that is within the normal range for the laboratory at the study center (or documentation of clinical insignificance in the subject's medical record by the investigator if outside the normal range) and measured ≤ 30 days prior to the date of surgery.
* History of inadequate response, contraindication, or refusal to medical therapy.

Exclusion Criteria:

* Body Mass Index (BMI) ≥ 42.
* History of prostate cancer or current/suspected bladder cancer.
* Prostate cancer should be ruled out before participation to the satisfaction of the investigator if Prostate-Specific Antigen (PSA) is above acceptable thresholds.
* Subjects with a history of actively treated bladder cancer within the past two (2) years.
* Bladder calculus or clinically significant bladder diverticulum (e.g., pouch size >20% of full bladder size).
* Active infection, including urinary tract infection.
* Prostatitis treated with antibiotics within 1 year of enrollment.
* Ever been diagnosed with a urethral stricture, meatal stenosis, or bladder neck contracture.
* Subject has damage to external urinary sphincter .
* Subject has diagnosis of stress urinary incontinence that requires treatment or daily pad or device use.
* Post-Void Residual (PVR) > 300 mL.
* Urinary retention at time of enrollment or subject has been catheterized in the 14 days prior to the surgical procedure.
* Subject has a history of intermittent self-catheterization.
* Previous prostate surgery or history of other lower urinary tract surgery such as e.g. urinary diversion, artificial urinary sphincter or penile prosthesis.
* Subjects on anticoagulants (if medication cannot be stopped before and after procedure) or known coagulopathy (except aspirin below 100mg/d).
* Any severe illness that would prevent complete study participation or confound study results.
* Participants using systematic immune-suppressants including corticosteroids; unable to withhold non-steroidal anti-inflammatory agents (Nonsteroidal anti-inflammatory drugs (NSAIDs), including aspirin) for 3-5 days prior to treatment except for low dose aspirin (e.g. less than or equal to 100mg).
* Participants using anticholinergics specifically for bladder problems. Use of medications with anticholinergic properties is allowable provided the patient does not have documented adverse urinary side effects from these medications.
* Contraindication to general or spinal anesthesia.
* Subject has any other disease or condition(s) that would interfere with completion of the study and follow up assessments, would increase risks of the procedure, or in the judgment of the investigator would potentially interfere with compliance to this study or would adversely affect outcomes.
* Subject is unwilling to accept a transfusion should one be required.

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2015-10-30 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2021-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gilling, M.D., Principal Investigator — Urology BOP; Claus Roehrborn, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (17):
- United States (12):
  - Urology Centers of Alabama, Birmingham, Alabama
  - San Diego Clinical Trials, La Mesa, California
  - University of Southern California, Institute of Urology, Los Angeles, California
  - Urology Associates, P.C., Englewood, Colorado
  - Adult & Pediatric Urology P.C., Omaha, Nebraska
  - Albany Medical College, Albany, New York
  - Weill Cornell Medical College, New York, New York
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - Houston Metro Urology, Houston, Texas
  - University of Vermont College of Medicine, Burlington, Vermont
  - Virginia Urology, Richmond, Virginia
- Royal Melbourne Hospital, Melbourne, Victoria, Australia
- Tauranga Urology Research Ltd., Tauranga, New Zealand
- United Kingdom (3):
  - Frimley Park Hospital, Frimley, Surrey
  - Princess of Wales Hospital, Bridgend, Wales
  - Addenbrooke's Treatment Center, Cambridge

REFERENCES:
- [Background] Gilling P, Barber N, Bidair M, Anderson P, Sutton M, Aho T, Kramolowsky E, Thomas A, Cowan B, Kaufman RP Jr, Trainer A, Arther A, Badlani G, Plante M, Desai M, Doumanian L, Te AE, DeGuenther M, Roehrborn C. WATER: A Double-Blind, Randomized, Controlled Trial of Aquablation(R) vs Transurethral Resection of the Prostate in Benign Prostatic Hyperplasia. J Urol. 2018 May;199(5):1252-1261. doi: 10.1016/j.juro.2017.12.065. Epub 2018 Jan 31. PMID 29360529
- [Background] Gilling PJ, Barber N, Bidair M, Anderson P, Sutton M, Aho T, Kramolowsky E, Thomas A, Cowan B, Roehrborn C. Randomized Controlled Trial of Aquablation versus Transurethral Resection of the Prostate in Benign Prostatic Hyperplasia: One-year Outcomes. Urology. 2019 Mar;125:169-173. doi: 10.1016/j.urology.2018.12.002. Epub 2018 Dec 12. PMID 30552937
- [Background] Gilling P, Barber N, Bidair M, Anderson P, Sutton M, Aho T, Kramolowsky E, Thomas A, Cowan B, Kaufman RP Jr, Trainer A, Arther A, Badlani G, Plante M, Desai M, Doumanian L, Te AE, DeGuenther M, Roehrborn C. Two-Year Outcomes After Aquablation Compared to TURP: Efficacy and Ejaculatory Improvements Sustained. Adv Ther. 2019 Jun;36(6):1326-1336. doi: 10.1007/s12325-019-00952-3. Epub 2019 Apr 26. PMID 31028614
- [Background] Gilling P, Barber N, Bidair M, Anderson P, Sutton M, Aho T, Kramolowsky E, Thomas A, Cowan B, Kaufman RP Jr, Trainer A, Arther A, Badlani G, Plante M, Desai M, Doumanian L, Te AE, DeGuenther M, Roehrborn C. Three-year outcomes after Aquablation therapy compared to TURP: results from a blinded randomized trial. Can J Urol. 2020 Feb;27(1):10072-10079. PMID 32065861
- [Background] Gilling PJ, Barber N, Bidair M, Anderson P, Sutton M, Aho T, Kramolowsky E, Thomas A, Kaufman RP Jr, Badlani G, Plante M, Desai M, Doumanian L, Te AE, Roehrborn CG. Five-year outcomes for Aquablation therapy compared to TURP: results from a double-blind, randomized trial in men with LUTS due to BPH. Can J Urol. 2022 Feb;29(1):10960-10968. PMID 35150215
- [Derived] Pimentel MA, Yassaie O, Gilling P. Urodynamic Outcomes After Aquablation. Urology. 2019 Apr;126:165-170. doi: 10.1016/j.urology.2019.01.020. Epub 2019 Feb 2. PMID 30721737
- [Derived] Chughtai B, Thomas D. Pooled Aquablation Results for American Men with Lower Urinary Tract Symptoms due to Benign Prostatic Hyperplasia in Large Prostates (60-150 cc). Adv Ther. 2018 Jun;35(6):832-838. doi: 10.1007/s12325-018-0722-0. Epub 2018 Jun 5. PMID 29873008

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: AQUABEAM System
  The AQUABEAM system, a personalized image-guided tissue removal system, utilizes proprietary heat-free high-velocity waterjet technology to resect and remove prostate tissue.
- Active Comparator: Transurethral Resection of the Prostate (TURP)
  Transurethral resection of the prostate (TURP) is a type of prostate surgery done to relieve moderate to severe urinary symptoms caused by an enlarged prostate, a condition known as benign prostatic hyperplasia (BPH)
Period: Treatment
Arm/Group | Treatment | Active Comparator
Started | 116 | 65
Completed | 116 | 65
Not Completed | 0 | 0
Period: 1 Week Follow-Up
Arm/Group | Treatment | Active Comparator
Started | 116 | 65
Completed | 116 | 65
Not Completed | 0 | 0
Period: 1 Month Follow-Up
Arm/Group | Treatment | Active Comparator
Started | 116 | 65
Completed | 116 | 65
Not Completed | 0 | 0
Period: 3 Months Follow-Up
Arm/Group | Treatment | Active Comparator
Started | 116 | 65
Completed | 116 | 65
Not Completed | 0 | 0
Period: 6 Months Follow-Up
Arm/Group | Treatment | Active Comparator
Started | 116 | 65
Completed | 116 | 63
Not Completed | 0 | 2
Period: 12 Months Follow-Up
Arm/Group | Treatment | Active Comparator
Started | 116 | 63
Completed | 115 | 61
Not Completed | 1 | 2
Period: 24 Months Follow-Up
Arm/Group | Treatment | Active Comparator
Started | 115 | 61
Completed | 112 | 60
Not Completed | 3 | 1
Period: 36 Months Follow-Up
Arm/Group | Treatment | Active Comparator
Started | 112 | 60
Completed | 97 | 55
Not Completed | 15 | 5
Period: 60 Months Follow-Up
Arm/Group | Treatment | Active Comparator
Started | 97 | 55
Completed | 58 | 32
Not Completed | 39 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Active Comparator | Total
Number analyzed (Participants) | 117 | 67 | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (7.3) | 65.8 (7.2) | 65.9 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 117 | 67 | 184
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 114 | 64 | 178
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 2 | 5
  Hispanic | 2 | 3 | 5
  Black | 2 | 2 | 4
  White | 109 | 59 | 168
  Other | 1 | 0 | 1
  NA | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 11 | 9 | 20
  United States | 61 | 32 | 93
  United Kingdom | 32 | 18 | 50
  Australia | 13 | 8 | 21

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Adverse Events (Clavien-Dindo Grading System Grade 2 or Higher or Any Grade 1 Event Resulting in Persistent Disability)
Description: The primary safety endpoint is the proportion of subjects with adverse events rated as probably or definitely related to the study procedure classified as Clavien-Dindo Grade 2 or higher or any Grade 1 event resulting in persistent disability (e.g. ejaculatory disorder or erectile dysfunction) evidenced through 3 months post treatment. Note that the Clavien-Dindo classification scheme is for grading postoperative complications not events that reflect lack of effective treatment. Results are presented as a percentage rounded to the whole number.
Time Frame: Three months post-treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment | Active Comparator
Number analyzed (Participants) | 116 | 65
percentage of participants | 26 [18.2 to 34.8] | 42 [29.4 to 54.4]

2. Primary Outcome: Change Score of IPSS Questionnaire Between Baseline and 6 Months
Description: The primary effectiveness endpoint is the IPSS change score from baseline to 6 months.
  International Prostate Symptom Score (IPSS) ranges from 0 to 35. A higher score indicates a worse outcome.
Time Frame: Six months post-treatment
Population: The variation between the overall number of participants analyzed for this outcome and the completed number on the participant flow at this follow-up is due to this specific outcome assessment not being done by all participants who completed this follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Active Comparator
Number analyzed (Participants) | 114 | 62
score on a scale | -16.9 (6.6) | -15.1 (7.9)

3. Other Pre Specified Outcome: Long-term Effectiveness as Measured by International Prostate Symptom Score (IPSS) at 60 Months
Description: Change score of International Prostate Symptom Score (IPSS) at 60 months as compared to baseline. Score range is from 0 to 35, with a low score associated with more favorable outcomes. Change score is calculated from two time points as the value at the 60 months point minus the value at the baseline.
Time Frame: 60 months following original surgical intervention
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Treatment | Active Comparator
Number analyzed (Participants) | 58 | 31
change in score on a scale | -15.1 (6.6) | -13.2 (8.2)

4. Other Pre Specified Outcome: International Prostate Symptom Score (IPSS) at 60 Months
Description: International Prostate Symptom Score (IPSS) at 60 months. Score range is from 0 to 35, with a low score associated with more favorable outcomes.
Time Frame: 60 months following original surgical intervention
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Treatment | Active Comparator
Number analyzed (Participants) | 58 | 31
score on a scale | 5.5 [1 to 28] | 6 [1 to 28]

5. Other Pre Specified Outcome: International Prostate Symptom Score Quality of Life (IPSS-QoL) at 60 Months
Description: International Prostate Symptom Score Quality of Life (IPSS-QoL) sub-score. Score range is from 0 to 6, with a low score associated with more favorable outcomes.
Time Frame: 60 months following original surgical intervention
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Active Comparator
Number analyzed (Participants) | 58 | 31
score on a scale | 1.6 (1.4) | 1.6 (1.5)

6. Other Pre Specified Outcome: Change in Maximum Urinary Flow Rate (Qmax) at 60 Months From Baseline
Description: Change in Uroflowmetry measurement of voided urine (in milliliters) per unit of time (in seconds) at 60 Months from Baseline. Change score is calculated from two time points as the value at the 60 months point minus the value at the baseline.
Time Frame: 60 months following original surgical intervention
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/s
Arm/Group | Treatment | Active Comparator
Number analyzed (Participants) | 41 | 26
mL/s | 8.7 (9.1) | 6.3 (7.5)

7. Other Pre Specified Outcome: Change in Post-void Residual (PVR) at 60 Months From Baseline
Description: Change in Post-void residual (PVR) urine test at 60 Months from Baseline. Change score is calculated from two time points as the value at the 60 months point minus the value at the baseline.
Time Frame: 60 months following original surgical intervention
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Treatment | Active Comparator
Number analyzed (Participants) | 41 | 25
mL | -62 (86) | -82 (94)

ADVERSE EVENTS:
Time Frame: 5 years
Description: There were no device-related adverse events reported in the study, and there were no unanticipated procedure-related adverse events reported in the study. Of the adverse events resulting in mortality, none were procedure-related, device-related, or urological.
Arm/Group | Treatment | Active Comparator
All-Cause Mortality (participants affected / at risk) | 4/116 | 1/65
Serious Adverse Events (participants affected / at risk) | 24/116 | 14/65
Other Adverse Events (participants affected / at risk) | 75/116 | 53/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=116) | Active Comparator (N=65)
Bladder neck contracture (non-procedure-related) (Renal and urinary disorders) | 1 | 1
Bleeding (Renal and urinary disorders) | 4 | 4
Cardiac (non-procedure-related) (Cardiac disorders) | 4 | 2
Non-urologic (General disorders) | 3 | 0
Other bleeding (non-procedure-related) (General disorders) | 2 | 0
Pain (Renal and urinary disorders) | 1 | 0
Penial infection (non-procedure-related) (Infections and infestations) | 0 | 1
Prostate cancer (non-procedure-related) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Stricture or adhesions (Renal and urinary disorders) | 1 | 1
Stricture or adhesions (non-procedure-related) (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 3 | 2
Urinary retention (non-procedure-related) (Renal and urinary disorders) | 0 | 1
Urinary tract infection (non-procedure-related) (Renal and urinary disorders) | 2 | 0
Urinary tract stones (non-procedure-related) (Renal and urinary disorders) | 1 | 1
Urinary urgency/frequency/difficulty/leakage (Renal and urinary disorders) | 1 | 0
Urinary urgency/frequency/difficulty/leakage (non-procedure-related) (Renal and urinary disorders) | 5 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=116) | Active Comparator (N=65)
Atrial fibrillation (non-procedure-related) (Cardiac disorders) | 1 | 1
Bladder neck contracture (Renal and urinary disorders) | 0 | 1
Bladder neck contracture (non-procedure-related) (Renal and urinary disorders) | 1 | 1
Bladder pain/spasm (Renal and urinary disorders) | 7 | 3
Bleeding (Renal and urinary disorders) | 12 | 6
Bleeding (non-procedure-related) (Renal and urinary disorders) | 5 | 5
Decreased libido (Reproductive system and breast disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 14 | 6
Dysuria (non-procedure-related) (Renal and urinary disorders) | 4 | 1
Erectile Dysfunction (Reproductive system and breast disorders) | 0 | 1
Erectile Dysfunction (non-procedure-related) (Reproductive system and breast disorders) | 7 | 6
Hydrocele (Renal and urinary disorders) | 0 | 1
Hypertension (non-procedure-related) (Cardiac disorders) | 3 | 2
Hypotension (Cardiac disorders) | 3 | 0
Non-urologic (General disorders) | 16 | 7
Overactive bladder (non-procedure-related) (Renal and urinary disorders) | 5 | 0
Pain (Renal and urinary disorders) | 8 | 4
Pain (non-procedure-related) (Renal and urinary disorders) | 2 | 1
Penile disorder (non-procedure-related) (Renal and urinary disorders) | 2 | 0
Perineal swelling (Renal and urinary disorders) | 0 | 1
Prostatitis (non-procedure-related) (Infections and infestations) | 2 | 2
Retrograde ejaculation (Reproductive system and breast disorders) | 8 | 16
Retrograde ejaculation (non-procedure-related) (Reproductive system and breast disorders) | 5 | 4
Rising PSA (non-procedure-related) (Renal and urinary disorders) | 4 | 1
Sexual dysfunction (non-procedure-related) (Reproductive system and breast disorders) | 0 | 1
Stricture or adhesions (Renal and urinary disorders) | 2 | 1
Stricture or adhesions (non-procedure-related) (Renal and urinary disorders) | 1 | 2
Swollen Testicles (Renal and urinary disorders) | 0 | 1
Urethral damage (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 8 | 3
Urinary retention (non-procedure-related) (Renal and urinary disorders) | 4 | 5
Urinary tract infection (Renal and urinary disorders) | 11 | 5
Urinary tract infection (non-procedure-related) (Renal and urinary disorders) | 6 | 4
Urinary tract stones (non-procedure-related) (Renal and urinary disorders) | 2 | 1
Urinary urgency/frequency/difficulty/leakage (Renal and urinary disorders) | 9 | 9
Urinary urgency/frequency/difficulty/leakage (non-procedure-related) (Renal and urinary disorders) | 18 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT02505919/Prot_002.pdf
  • Statistical Analysis Plan (2016-09-23): https://cdn.clinicaltrials.gov/large-docs/19/NCT02505919/SAP_001.pdf